CLINICAL TRIAL: NCT01222702
Title: A Multi-center, Double-blind, Randomized, Active Reference, Parallel Group Study to Evaluate the Efficacy, Safety and Tolerability of a 10-day Twice Daily Oral Administration of Three Doses of Cadazolid (ACT-179811) in Subjects With Clostridium Difficile Associated Diarrhea (CDAD)
Brief Title: Efficacy, Safety and Tolerability of Cadazolid in Subjects With Clostridium Difficile Associated Diarrhea (CDAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-061A201
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Clostridium Difficile Infection
Keywords: CDIFF; CDAD; CDI; Clostridium difficile infection
MeSH Terms: conditions — Clostridium Infections | interventions — cadazolid; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cadazolid 250 mg (Experimental): Subjects received 250 mg of reconstituted cadazolid suspension twice daily and one placebo-matching vancomycin capsule four times daily for 10 days
  Interventions: Drug: Cadazolid; Drug: Placebo-matching vancomycin
- Cadazolid 500 mg (Experimental): Subjects received 500 mg of reconstituted cadazolid suspension twice daily and one placebo-matching vancomycin capsule four times daily for 10 days
  Interventions: Drug: Cadazolid; Drug: Placebo-matching vancomycin
- Cadazolid 1000 mg (Experimental): Subjects received 1000 mg of reconstituted cadazolid suspension twice daily and one placebo-matching vancomycin capsule four times daily for 10 days
  Interventions: Drug: Cadazolid; Drug: Placebo-matching vancomycin
- Vancomycin 125 mg (Active Comparator): Subjects received one vancomycin capsule (125 mg) four times daily and reconstituted placebo-matching cadazolid suspension twice daily for 10 days
  Interventions: Drug: Vancomycin; Drug: Placebo-matching cadazolid

INTERVENTIONS:
Drug: Cadazolid — Cadazolid, provided as powder (250 mg, 500 mg or 1000 mg) to be reconstituted as a suspension prior to oral administration
  Other Names: ACT-179811
  Arms: Cadazolid 1000 mg; Cadazolid 250 mg; Cadazolid 500 mg
Drug: Vancomycin — Vancomycin, provided as capsules (125 mg) for oral administration
  Other Names: Vancomycin hydrochloride
  Arms: Vancomycin 125 mg
Drug: Placebo-matching cadazolid — Placebo of cadazolid powder for oral suspension
  Arms: Vancomycin 125 mg
Drug: Placebo-matching vancomycin — Placebo of vancomycin capsules
  Arms: Cadazolid 1000 mg; Cadazolid 250 mg; Cadazolid 500 mg

SUMMARY:
Cadazolid is a new antibiotic developed for the treatment of Clostridiun difficile associated diarrhea (CDAD), also known as Clostridium Difficile Infection (CDI). The purpose of the study was to evaluate the efficacy and safety of different doses of cadazolid in order to find the dose of cadazolid to be used for further clinical development of the compound in subjects with CDAD.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female
* At least 18 years of age
* With a diagnosis of Clostridium Difficile-associated diarrhea (CDAD): first occurrence or first recurrence.

Key Exclusion Criteria:

* Concurrent life threatening condition.
* Immuno-compromised subjects, concomittant immuno-suppresive treatment.
* Concomitant antimicrobial treatment for CDAD.
* Any circumstances or conditions, which, in the opinion of the investigator, would affect full participation of the subject in the study or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-01-25 (Actual); Primary Completion 2012-10-16 (Actual); Study Completion 2012-11-12 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate at test-of-cure | Day 13 or 24-72 hours after end of treatment
  Percentages of subjects with clinical cure are calculated, with clinical cure being defined as resolution of diarrhea with no further Clostridium Difficile-associated diarrhea (CDAD) treatment required at test-of-cure (TOC) visit.
  Resolution of diarrhea was defined as the occurrence of ≤ 2 semi-formed or formed stools during 24 h for at least 2 consecutive 24 h periods.

SECONDARY OUTCOMES:
Recurrence rate | Between Day 13 and Day 41 (within 4 weeks after end of treatment)
  Percentages of subjects with recurrence are calculated, with recurrence being defined as the occurrence of diarrhea (> 3 liquid or unformed stools within 24 h associated with positive C. difficile toxin A/B assay) within 4 weeks after EOT in subjects clinically cured (at test-of-cure).
Sustained cure rate | Between Day 13 and day 41 (within 4 weeks after end of treatment)
  Percentages of subjects with sustained cure are calculated, with sustained cure being defined as clinical cure without CDAD recurrence up to the end of study
Time to resolution of diarrhea | From Day 1 up to Day 13 (or 24-72 hours after end of treatment)
  Time to resolution of diarrhea was defined as the time (h) from the first intake of study treatment to the time (occurrence) of the first stool meeting the criteria for resolution of diarrhea up to test-of-cure.
Incidence of treatment-emergent adverse events | From Day 1 to Day 14
  Percentage of subjects with any adverse events in each group from first study treatment intake up to 3 days after last study drug intake
Adverse events leading to premature discontinuation of study treatment | Up to Day 10
  Number of patients in each group who discontinued the study treatment due to an adverse event

OTHER OUTCOMES:
Modified clinical cure rate | Day 13 or 24-72 hours after end of treatment
  Percentage of subjects with modified clinical cure (mCC) is reported, with mCC defined as the occurrence of ≤ 3 liquid or unformed stools and any number of semi-formed or formed stools per day for at least two consecutive days, and thereafter maintained up to TOC visit. In addition, no concomitant medication active against CDAD received from the start of study treatment up to TOC

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Charef, DVM, Study Director — Actelion
Locations (23):
- United States (11):
  - Clinical Investigative Site 6902, Newark, Delaware
  - Clinical Investigative Site 6919, Jacksonville, Florida
  - Clinical Investigative Site 6938, Orlando, Florida
  - Clinical Investigative Site 6930, Decatur, Georgia
  - Clinical Investigative Site 6935, Marietta, Georgia
  - Clinical Investigative Site 6915, Idaho Falls, Idaho
  - Clinical Investigative Site 6906, Chicago, Illinois
  - Clinical Investigative Site 6917, Boston, Massachusetts
  - Clinical Investigative Site 6936, Royal Oak, Michigan
  - Clinical Investigative Site 6903, Columbus, Ohio
  - Clinical Investigative Site 6914, Houston, Texas
- Canada (4):
  - Clinical Investigative Site 6605, Victoria, British Columbia
  - Clinical Investigative Site 6601, Montreal, Quebec
  - Clinical Investigative Site 6606, Sherbrooke, Quebec
  - Clinical Ivestigative Site 6602, Calgary
- Germany (3):
  - Clinical Investigative Site 6632, Cologne
  - Clinical Investigative Site 6633, Regensburg
  - Clinical Investigative Site 6634, Ulm
- Italy (2):
  - Clinical Investigative Site 6734, Busto Arsizio
  - Clinical Investigative Site 6735, Modena
- Clinical Investigative Site 6702, Örebro, Sweden
- United Kingdom (2):
  - Clinical Investigative Site 6801, Blackpool
  - Clinical Investigative Site 6804, York

REFERENCES:
- [Result] Louie T, Nord CE, Talbot GH, Wilcox M, Gerding DN, Buitrago M, Kracker H, Charef P, Cornely OA. Multicenter, Double-Blind, Randomized, Phase 2 Study Evaluating the Novel Antibiotic Cadazolid in Patients with Clostridium difficile Infection. Antimicrob Agents Chemother. 2015 Oct;59(10):6266-73. doi: 10.1128/AAC.00504-15. Epub 2015 Jul 27. PMID 26248357
- [Result] Gerding DN, Hecht DW, Louie T, Nord CE, Talbot GH, Cornely OA, Buitrago M, Best E, Sambol S, Osmolski JR, Kracker H, Locher HH, Charef P, Wilcox M. Susceptibility of Clostridium difficile isolates from a Phase 2 clinical trial of cadazolid and vancomycin in C. difficile infection. J Antimicrob Chemother. 2016 Jan;71(1):213-9. doi: 10.1093/jac/dkv300. Epub 2015 Oct 3. PMID 26433782